CLINICAL TRIAL: NCT00845169
Title: The Role of Nitric Oxide Synthase Isoforms in the Cardiovascular Effects of Air Pollution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); Umeå University (Other)
Responsible Party: Principal Investigator, Jeremy Langrish, Clinical Lecturer and Specialty Registrar in Cardiology, University of Edinburgh
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: DNR 08-185M/2
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Endothelial Dysfunction
Keywords: Air Pollution; Nitric Oxide; Nitric Oxide Synthase; Diesel exhaust; endothelial dysfunction
MeSH Terms: interventions — omega-N-Methylarginine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diesel Exposure (Experimental): 1 hour exposure to diesel exhaust at 300 µg/m3 during intermittent exercise
  Interventions: Procedure: Forearm vascular study
- Air Exposure (Experimental): 1 hour exposure to filtered air during intermittent exercise
  Interventions: Procedure: Forearm vascular study

INTERVENTIONS:
Procedure: Forearm vascular study — Forearm venous occlusion plethysmography to measure forearm blood flow during intrabrachial infusion of nitric oxide synthase inhibitors L-NMMA (2-8 µg/min), S-methionyl-L-citrulline (25-200 nmol/min) and 1400W (100-1000 nmol/min) and positive control norepinephrine (60-540 pmol/min)
  Other Names: 1400W; SMTC; L-NMMA; Noreadrenaline; NorAd

SUMMARY:
Exposure to air pollution has been linked to increased cardiorespiratory morbidity and mortality. The exact component of air pollution that mediates this effect is unknown, but the link is strongest for fine combustion derived particulate matter derived from traffic sources. Recently, it has been demonstrated that inhalation of diesel exhaust impairs vascular vasomotor tone and endogenous fibrinolysis. The mechanism underlying these detrimental vascular is unclear, but is thought to be via oxidative stress and altered bioavailability of endogenous nitric oxide. In these studies we plan to elucidate the role of endogenous nitric oxide synthase isoforms (NO) in the adverse vascular responses observed following exposure to diesel exhaust.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Regular medication use (except oral contraceptive pill)
* Current smokers
* Significant occupational exposure to air pollution
* Intercurrent illness

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Forearm blood flow measured by venous occlusion plethysmography during intraarterial infusion of nitric oxide synthase inhibitors L-NMMA, SMTC and 1400W and positive control norepinephrine. | 2-4 hours after exposure

SECONDARY OUTCOMES:
Plasma nitrite concentration | During forearm study

CONTACTS AND LOCATIONS:
Overall Officials: Anders Blomberg, MD PhD, Principal Investigator — Umeå University; David E Newby, PhD FRCP, Principal Investigator — University of Edinburgh
Locations (1):
- Umeå University, Umeå, Sweden